CLINICAL TRIAL: NCT06006117
Title: Phase III, Multicenter, Open Label, Randomized, Controlled Study Investigating Mosunetuzumab-Lenalidomide Versus Investigator Choices in Patients With Relapsed or Refractory Marginal Zone Lymphoma
Brief Title: Mosunetuzumab-Lenalidomide Versus Investigator Choices in Patients With Relapsed or Refractory Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARSUN
Record Dates: First submitted 2023-07-27; First posted 2023-08-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-01

CONDITIONS: Marginal Zone Lymphoma
Keywords: Bispecific antibodies, Subcutaneous; Step-up dosing; Marginal Zone Lymphoma; Investigator choices; R/R MZL
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Bendamustine Hydrochloride; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Arm A - Experimental arm: Mosunetuzumab-Lenalidomide
  Arm B - Comparator arms (Investigator Choices):
  * Rituximab-Lenalidomide
  * Rituximab-Bendamustine
  * Rituximab-CHOP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Mosunetuzumab and Lenalidomide (Experimental): * Mosunetuzumab will be administered SC (21 days first cycle, then 28 days next cycles)
    * C1 (21-days cycle): step-up dosing schedule 5 mg Day 1, 45 mg on Day 8 and 45 mg Day 15
    * C2 to C12: 45 mg D1 28-days cycles
  * Lenalidomide PO starting dose is based on patient's creatinine clearance from Day 1 to Day 21 from cycles C2 to C6 (cycles of 28 days)
  Interventions: Drug: Mosunetuzumab (SC); Drug: Lenalidomide
- Arm 2: Rituximab-Lenalidomide (28-days cycles) (Active Comparator): * Rituximab* 375 mg/m2 intravenously at Day 1 cycle 1, and then subcutaneous (1400 mg, flat dose) at D1 of cycles 2-12
  * Lenalidomide PO starting dose is based on patient's creatinine clearance, D1-21 from cycle 1 to cycle 6
  Interventions: Drug: Rituximab (R); Drug: Lenalidomide
- Arm 3: Rituximab-Bendamustine (28-days cycles) (Active Comparator): * Rituximab* 375 mg/m2 intravenously at cycle 1 Day 1, and then subcutaneous (1400 mg, flat dose) at D1 of cycles 2 to 6** (28-days cycles) and then at D1 of three additional 56-days cycles (C7 to C9). **For patients in complete response (CR) at 3 cycles, if Bendamustine is stopped, then Rituximab should also be omitted for C5 and C6.
  * Bendamustine IV 70 or 90 mg/m² (according to the investigator's judgment) D1 and D2/28 days x 6 cycles 28 days cycles). For patients in complete response (CR) at 3 cycles, Bendamustine and Rituximab could be stopped after 4 cycles at investigator discretion
  Interventions: Drug: Rituximab (R); Drug: Bendamustine
- Arm 4: Rituximab-CHOP (21-days cycles) (Active Comparator): * Rituximab* 375 mg/m2 intravenously at Day 1 cycle 1, and then subcutaneous (1400 mg, flat dose) at D1 of cycles 2 to 6 (21-days cycles), and then at D1 of three additional 56-days cycles (C7 to C9)
  * CHOP, IV standard dose from cycle 1 to 6
  Interventions: Drug: Rituximab (R); Drug: CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone)

INTERVENTIONS:
Drug: Mosunetuzumab (SC) — ○ Mosunetuzumab will be administered SC (21 days first cycle, then 28 days next cycles)
  * C1 (21-days cycle): step-up dosing schedule 5 mg Day 1, 45 mg on Day 8 and 45 mg Day 15
  * C2 to C12: 45 mg D1 28-days cycles
  Other Names: Mosunetuzumab
  Arms: Arm 1: Mosunetuzumab and Lenalidomide
Drug: Rituximab (R) — Rituximab* 375 mg/m2 intravenously at Day 1 cycle 1, and then subcutaneous (1400 mg, flat dose) at D1 of cycles 2-12
  Other Names: Rituximab
  Arms: Arm 2: Rituximab-Lenalidomide (28-days cycles); Arm 3: Rituximab-Bendamustine (28-days cycles); Arm 4: Rituximab-CHOP (21-days cycles)
Drug: Bendamustine — ○ Bendamustine IV 70 or 90 mg/m² (according to the investigator's judgment) D1 and D2/28 days x 6 cycles 28 days cycles). For patients in complete response (CR) at 3 cycles, Bendamustine and Rituximab could be stopped after 4 cycles at investigator discretion
  Arms: Arm 3: Rituximab-Bendamustine (28-days cycles)
Drug: CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone) — CHOP, IV standard dose from cycle 1 to 6
  Other Names: CHOP
  Arms: Arm 4: Rituximab-CHOP (21-days cycles)
Drug: Lenalidomide — Cycles 2 to 6 (28-day cycles): starting dose is based on patient's creatinine clearance, from day 1 to day 21, once a day, rest period from day 22 to day 28
  Arms: Arm 1: Mosunetuzumab and Lenalidomide; Arm 2: Rituximab-Lenalidomide (28-days cycles)

SUMMARY:
This is an open label, multi-center, international, randomized phase III trial to compare the efficacy of Mosunetuzumab-Lenalidomide with investigator choices exclusively in R/R MZL patients. Patients with a proven diagnosis of EMZL, SMZL or NMZL subtypes and previously treated with at least one prior systemic treatment and not more than three prior lines are eligible. Previous treatment line must include at least one systemic line with a drug targeting CD20 (monoclonal antibody at least 2 cycles) with or without chemotherapy (R-CHOP, R-Bendamustine, R-CVP, R-Chlorambucil at least 2 cycles) or targeted treatment such as Ibrutinib.

The patients will be Randomized as follows:

Arm A - Experimental arm:

• Mosunetuzumab-Lenalidomide

Arm B - Comparator arms ( Investigator Choices):

* Rituximab-Lenalidomide
* Rituximab-Bendamustine
* Rituximab-CHOP

DETAILED DESCRIPTION:
This is an open label, multi-center, international, randomized phase III trial to compare the efficacy of Mosunetuzumab-Lenalidomide with investigator choices exclusively in R/R MZL patients. Patients with a proven diagnosis of EMZL, SMZL or NMZL subtypes and previously treated with at least one prior systemic treatment and not more than three prior lines are eligible. Previous treatment line must include at least one systemic line with a drug targeting CD20 (monoclonal antibody at least 2 cycles) with or without chemotherapy (R-CHOP, R-Bendamustine, R-CVP, R-Chlorambucil at least 2 cycles) or targeted treatment such as Ibrutinib.

Patients are stratified according to MZL subtypes and time to progression of disease after first-line within 2 years (POD24) < 2 years or > 2 years.

Mosunetuzumab will be administered sub-cutaneously (SC) (21 days first cycle, then 28 days next cycles) and Lenalidomide will be given PO 20 mg/day from Day 1 to Day 21 from cycles C2 to C6. For each patient, investigator choice had to be decided before randomization between Rituximab-Lenalidomide and Rituximab-chemotherapy (R-Bendamustine or R-CHOP).

The primary efficacy endpoint for comparison is the Progression-free survival (PFS) as determined by investigator (Lugano criteria 2014). Secondary objectives include CR24 as determined by investigator (at 24 months) according to Lugano criteria 2014 and by central review based on PET result, Overall response rate (ORR) and CR other than CR24 as determined by investigator, or by central review based on PET result according to Lugano Criteria 2014. 260 patients are planned to be enrolled in France, Belgium, Germany, Italy and Portugal

ELIGIBILITY:
Inclusion criteria:

1. Have a diagnosis of MZL, of extranodal (EMZL) or splenic (SMZL based on the Matutes score and CD20 + CD11c + CD180 + CD43 + CD200 expression and validated by a centralized review) or nodals (NMZL) subtypes. In case of large dissemination, disseminated MZL (as evaluated by investigator; please contact the Sponsor to discuss any doubt) will be included as DMZL and included in NMZL subtype.
2. Have been treated with at least one prior systemic treatment and not more than three prior lines. Previous line must include at least one systemic line with a drug targeting CD20 (monoclonal antibody at least 2 cycles; patient treated with monoclonal antibody monotherapy should have received at least 4 weekly injections) with or without chemotherapy (R-CHOP, R-Bendamustine, R-CVP, R-Chlorambucil at least 2 cycles) or targeted treatment such as Ibrutinib (at least 1 month). Patients previously treated by lenalidomide are eligible if the last administration of lenalidomide is superior to 12 months before C1D1. When randomized in comparator arm, those patients should require R-chemo. Prior local therapy (including surgery, radiotherapy antibiotics for H. pylori-positive gastric lymphoma, and antiviral for hepatitis C virus) is not considered as one line of treatment
3. Signed Informed Consent Form
4. Age ≥ 18 years at the time of signing the informed consent form
5. Ability to comply with the study protocol and procedures and required hospitalizations, in the investigator's judgement
6. Eastern Cooperative Oncology Group (ECOG) performance score (PS) of ≤ 2
7. Have a symptomatic disease requiring a systemic treatment
8. Not eligible for a local treatment including radiotherapy or surgery
9. Stage I disease of EMZL, SMZL or NMZL may be eligible only if not candidate to local therapy (surgery or radiotherapy).
10. Measurable disease in at least two perpendicular dimensions on an imaging scan is defined as: lymph node or nodal mass bi-dimensional measurement with ≥ 15 mm in longest transverse diameter or the short diameter must measure ≥ 10 mm regardless of the longest transverse diameter.

    Spleen is considered as a measurable disease if vertical axis is higher than 13 cm.
11. Adequate hematopoietic function at screening as follows unless cytopenia is clearly due to marrow involvement of MZL or hypersplenism or autoimmune thrombocytopenia:

    11.1. Platelet count ≥ 75 G/L; in cases of thrombocytopenia clearly due to marrow involvement of MZL or hypersplenism or auto-immune thrombocytopenia, platelet count should be ≥ 30 G/L Washout platelet transfusion is 7 days between transfusion and D1 of starting treatment

    11.2. ANC ≥ 1 G/L unless neutropenia is clearly due to marrow involvement of MZL or hypersplenism. G-CSF is not allowed within 7 days before starting treatment

    11.3. Total hemoglobin ≥ 8 g/dL unless anemia is clearly due to marrow involvement of MZL or hypersplenism or autoimmune hemolytic anemia. Washout erythrocyte transfusion is 7 days between transfusion and D1 of starting treatment
12. Serum total bilirubin ≤ 1.5 x the upper limit of normal (ULN) (or ≤3 x ULN for patients with Gilbert syndrome),
13. AST or ALT ≤ 2.5 x ULN, unless directly attributable to the patient's MZL
14. Measured or estimated creatinine clearance ≥ 40 mL/min by institutional standard method
15. Patients who are hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (HBcAb) positive, must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation. Patients who are hepatitis B surface antigen (HBsAg) negative, hepatitis B surface antibody (anti-HBsAb) positive and hepatitis B core antibody (HBcAb) negative are eligible,
16. Contraception:

    16.1. For women of childbearing potential (WOCBP): Serum test pregnancy at screening and Day 1 before first dose. And then monthly until end of chemotherapy or end of lenalidomide. Efficient contraceptive method is required during the treatment period (including periods of treatment interruption), for at least 28 days after the final dose of lenalidomide (if applicable), 3 months after the final dose of mosunetuzumab and tocilizumab (if applicable), 12 months after the final dose of CHOP (if applicable), 6 months after the final dose of bendamustine (if applicable) and 12 months after the final dose of rituximab (if applicable).

    16.2. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period (including periods of treatment interruption), and for at least 28 days after the final dose of lenalidomide (if applicable), 2 months after the final dose of tocilizumab (if applicable), 6 months after the final dose of CHOP (if applicable), 3 months after the final dose of bendamustine and 12 months after the final dose of rituximab (if applicable).
17. Patient covered by any social security system (France).
18. Patient who understands and speak one of the country official languages.

Exclusion criteria:

1. MZL with histologic transformation to high-grade lymphoma
2. Participants who have received any of the following treatments prior to study entry:

   * Treatment with mosunetuzumab or other CD20/CD3-directed bispecific antibodies
   * Allogeneic stem cell transplant
3. Participants who have received any of the following treatments, whether investigational or approved, within the respective time periods prior to initiation of study treatment:

   * Radiotherapy within 2 weeks prior to the first dose of study treatment
   * Autologous stem cell transplant within 100 days prior to first study treatment
   * Use of monoclonal antibodies within 4 weeks prior to first study treatment
   * Systemic immunosuppressive medications (including, but not limited to, Cyclophosphamide, Azathioprine, Methotrexate, Thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to first dose of study treatment (C1D1); Systemic corticosteroid treatment <20 mg/day Prednisone or equivalent and inhaled corticosteroids are permitted. Last dose of corticosteroid ≥20 mg/day Prednisone or equivalent will not be permitted during the last 15 days before inclusion.

   Administration of acute, low-dose, systemic immunosuppressant medications (e.g., single dose of 4 mg/day of dexamethasone for nausea or B-symptoms) is permitted during 4 days without washout.

   - Any other anti-cancer investigational therapy within 4 weeks prior to initiation of study treatment.
4. Pregnant or breastfeeding or intending to become pregnant during the study or within 28 days after the final dose of lenalidomide, 3 months after the final dose of mosunetuzumab and tocilizumab (if applicable), 12 months after the final dose of CHOP, 6 months after the final dose of bendamustine and 12 months after the final dose of rituximab (if applicable). Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment.
5. Received a live, attenuated vaccine within 4 weeks before first dose of study treatment, or in whom it is anticipated that such a live attenuated vaccine will be required during the study period or within 5 months after the final dose of study treatment, except for acute pandemic situation such COVID19
6. Active or history of CNS lymphoma or leptomeningeal infiltration
7. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody therapy (or recombinant antibody-related fusion proteins) - grade 3 and 4
8. Known hypersensitivity to biopharmaceuticals produced in CHO cells or any component of the mosunetuzumab, rituximab, tocilizumab, lenalidomide, or thalidomide formulation, including Mannitol
9. Patients unable to receive adequate prophylaxis and/or therapy for thromboembolic events (aspirin or low molecular weight heparin)
10. History of prior malignancy, except for conditions as listed below if patients have recovered from the acute side effects incurred as a result of previous therapy:

    * Malignancies treated with curative intent and with no known active disease present for ≥ 2 years before enrollment
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated cervical carcinoma in situ without evidence of disease
    * Surgically/adequately treated low grade, early stage I, localized prostate in situ carcinoma
11. Participants with infections requiring IV treatment with antibiotics or hospitalization (Grade 3 or 4) within the last 4 weeks prior to inclusion or known active bacterial, viral (including SARS-CoV-2), fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds),
12. Evidence of any significant, concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to:

    * Significant cardiovascular disease [e.g., Objective Class C or D heart diseases (cf. Classes of Heart Failure | American Heart Association)], myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina)
    * Significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
    * Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis
    * Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 1 year and have no residual neurologic deficits as judged by the investigator are allowed. Participants with a history of epilepsy who have had no seizures in the past 2 years with or without anti-epileptic medications can be eligible.
13. History of confirmed progressive multifocal leukoencephalopathy (PML)
14. Known Positive serologic HIV test at screening
15. Acute or chronic hepatitis C virus (HCV) infection Participants who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation.
16. Known or suspected history of hemophagocytic lymphohistiocytosis
17. Known or suspected chronic active Epstein-Barr virus (EBV) infection within the last 4 weeks prior to inclusion
18. History of erythema multiforme, Grade ≥3 rash, or blistering following prior treatment with immunomodulatory derivatives
19. History of interstitial lung disease (ILD), drug-induced pneumonitis, and autoimmune pneumonitis
20. Active autoimmune disease requiring treatment
21. History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis; except:

    * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with a history of disease-related immune thrombocytopenic purpura or autoimmune hemolytic anemia may be eligible.
    * Patients with a remote history of, or well-controlled autoimmune disease, with a treatment-free interval from immunosuppressive therapy for 12 months may be eligible after review and discussion with the Medical Monitor.
22. Recent major surgery with risk of bleeding within 4 weeks prior to first study treatment administration (C1D1)
23. History of solid organ transplantation
24. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes an individual's safe participation in and completion of the study
25. Person deprived of his/her liberty by a judicial or administrative decision
26. Person hospitalized without consent
27. Adult person under legal protection
28. Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness
29. patient unable to receive at least one of the three regimens of the comparator arm (ICT). As in usual practice, physician has to verify the absence of contraindication to the use of the drugs, hypersensitivity, and to take into account the lymphoma history and previous treatment scheme used
30. Suspicion or clinical evidence of transformed lymphoma at enrollment by investigator assessment (e.g. very high SUV (regarding SUV of other lesions) in at least one lesion that was not biopsied, and discordant with SUV of biopsied lesion, LDH > 2.5 ULN in a context of rapidly progressive disease, etc. (Please contact the Sponsor to discuss any possible inclusion in borderline cases or any doubt).
31. Uncontrolled symptomatic pleural or serous effusion requiring urgent treatment within 48 hours (patients with controlled disease after adequate pleural/serous drainage and/or effective pleurX™ or similar system are eligible).
32. Uncontrolled symptomatic ureterohydronephrosis resulting in renal failure (patients with adequate management i.e. ureteral catheter or double J stent allowing renal failure control are eligible).
33. MZL with high tumor burden defined as:

    * Lymphocytes ≥ 25 G/L, and/or
    * Spleen ≥ 17 cm of greatest axis, and/or
    * Lymph nodes ≥ 10 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as determined by investigator | After 122 events = approximately 4.5 years and after 163 events = approximately 6.5 years (event = progression or death)
  according to Lugano criteria 2014

SECONDARY OUTCOMES:
Complete Response rate (CR) as determined by investigator (CR24) | 2 years
  according to Lugano criteria 2014
Complete response rate (CR) by blinded central review (CR24) | 2 years
  based on PET result according to Lugano Criteria 2014
Overall response rate (ORR) as determined by investigator | 6 months for patients with Mosunetuzumab-Lenalidomide, Rituximab-Lenalidomide or R-CHOP, 3 months for patients with Rituximab-bendamustine
  according to Lugano Criteria 2014
Overall response rate (ORR) as determined by investigator | 12 months
  according to Lugano Criteria 2014
Overall response rate (ORR) as determined by investigator | 24 months
  according to Lugano Criteria 2014
Overall response rate (ORR) as determined by investigator | 36 months
  according to Lugano Criteria 2014
Overall response rate (ORR) as determined by investigator | 48 months
  according to Lugano Criteria 2014
Overall response rate (ORR) as determined by investigator | 60 months
  according to Lugano Criteria 2014
Overall response rate (ORR) by blinded central review | 6 months for patients with Mosunetuzumab-Lenalidomide, Rituximab-Lenalidomide or R-CHOP, 3 months for patients with Rituximab-bendamustine
  based on PET result according to Lugano Criteria 2014
Overall response rate (ORR) by blinded central review | 12 months
  based on PET result according to Lugano Criteria 2014
Overall response rate (ORR) by blinded central review | 24 months
  based on PET result according to Lugano Criteria 2014
Overall response rate (ORR) by blinded central review | 36 months
  based on PET result according to Lugano Criteria 2014
Overall response rate (ORR) by blinded central review | 48 months
  based on PET result according to Lugano Criteria 2014
Overall response rate (ORR) by blinded central review | 60 months
  based on PET result according to Lugano Criteria 2014
CR rate other than CR24 as determined by investigator | 6 months for patients with Mosunetuzumab-Lenalidomide, Rituximab-Lenalidomide or R-CHOP, 3 months for patients with Rituximab-bendamustine
  according to Lugano Criteria 2014
CR rate other than CR24 as determined by investigator | 12 months
  according to Lugano Criteria 2014
CR rate other than CR24 as determined by investigator | 24 months
  according to Lugano Criteria 2014
CR rate other than CR24 as determined by investigator | 36 months
  according to Lugano Criteria 2014
CR rate other than CR24 as determined by investigator | 48 months
  according to Lugano Criteria 2014
CR rate other than CR24 as determined by investigator | 60 months
  according to Lugano Criteria 2014
CR rate other than CR24 by blinded central review | 6 months for patients with Mosunetuzumab-Lenalidomide, Rituximab-Lenalidomide or R-CHOP, 3 months for patients with Rituximab-bendamustine
  based on PET result according to Lugano Criteria 2014
CR rate other than CR24 by blinded central review | 12 months
  based on PET result according to Lugano Criteria 2014
CR rate other than CR24 by blinded central review | 24 months
  based on PET result according to Lugano Criteria 2014
CR rate other than CR24 by blinded central review | 36 months
  based on PET result according to Lugano Criteria 2014
CR rate other than CR24 by blinded central review | 48 months
  based on PET result according to Lugano Criteria 2014
CR rate other than CR24 by blinded central review | 60 months
  based on PET result according to Lugano Criteria 2014
Duration of response (DOR) | 6.5 years
  time from the first occurrence of a documented objective response to progression/relapse or death from any cause
Event-free survival (EFS) | 6.5 years
  time from the date of randomization to the event of death of from any cause, disease progression or relapse, early discontinuation of the treatment because of any reason or first documented administration of any new anti-lymphoma treatment
Time to next anti-lymphoma treatment (TTNLT) | 6.5 years
  time from the date of randomization to the date of first documented administration of any new anti-lymphoma treatment
Histological transformation rate | 6.5 years
  percentage of transformation from MZL to diffuse large B-cell lymphoma
Safety: incidence and severity of Adverse Events (AE), of Serious Adverse Events (SAE), of Cytokine Release Syndrome (CRS), of AE grade 3 or 4 of study-drug_related events, incidence of Death and Secondary Primary Malignancies | 6.5 years
  Safety described according to actual treatment arm received
Tolerability : number of dose interruptions, dose reductions, and dose intensity, and study treatment discontinuation because of adverse events | 6.5 years
  Tolerability described according to actual treatment arm received
Health related quality of life as measured by the EQ-5D-5L | 7 months
  described by domains (Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression) and with the global score
Health related quality of life as measured by the EQ-5D-5L | 12 months
  described by domains (Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression) and with the global score
Health related quality of life as measured by the EQ-5D-5L | 24 months
  described by domains (Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression) and with the global score

CONTACTS AND LOCATIONS:
Overall Officials: Catherine THIEBLEMONT, Pr, Principal Investigator — Lymphoma Study Association; Sylvain CARRAS, Principal Investigator — Lymphoma Study Association
Locations (48):
- Belgium (4):
  - INSTITUT JULES BORDET - Service Hématologie, Anderlecht
  - UNIVERSITE CATHOLIQUE DE LOUVAIN SAINT-LUC - Service Hématologie, Brussels
  - UNIVERSITAIR ZIEKENHUIS GENT - Service Hématologie, Ghent
  - CHU UCL NAMUR - SITE GODINNE - Service Hématologie, Yvoir
- France (23):
  - CHU d'Amiens, Amiens
  - CH d'Avignon - Hopital Henri Duffaut, Avignon
  - CH de la Côte Basque - Hôpital de Bayonne, Bayonne
  - CHRU Besançon - Hôpital Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Chu Estaing, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble - Hôpital Albert Michallon, La Tronche
  - CHRU de LILLE - Claude Huriez, Lille
  - Institut Paoli Calmette, Marseille
  - CH Saint-Eloi, Montpellier
  - CHU de Nancy - Brabois, Nancy
  - Centre Catherine de Sienne, Nantes
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - CHR d'Orléans, Orléans
  - APHP - Hôpital Saint Louis, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
- Germany (9):
  - KLINIKUM ST. MARIEN AMBERG - Hämatologie/Onkologie, Amberg
  - Helios Klinikum Berlin-Buch - Klinik für Hämatologie und Stammzelltransplantation, Berlin
  - UNIVERSITAETSKLINIKUM SCHLESWIG-HOLSTEIN - Med. Klinik II - Hämatologie und Onkologie, Kiel
  - KLINIKUM DER STADT LUDWIGSHAFEN - Hämatologie, Ludwigshafen
  - UNIVERSITATSKLINIKUM REGENSBURG - Klinik für Innere Medizin III, Regensburg
  - ROBERT BOSCH KRANKENHAUS - Hämatologie, Onkologie und Palliativmedizin, Stuttgart
  - MUTTERHAUS DER BORROMAERINNEN - Hämatologie, Trier
  - UNIV KLINIKUM ULM - INNERE MEDIZIN III - Hämatologie, Ulm
  - UNIVERSITY WURZBURG - Hämatologie, Würzburg
- Italy (11):
  - POLICLINICO SANT'ORSOLA-MALPIGHI - Ematologia, Bologna
  - INSTITUTO ONCOLOGICO VENETO I.R.C.C.S - Ematologia, Castelfranco Veneto
  - AZIENDA OSPEDALIERA S. CROCE E CARLE CUNEO - Ematologia, Cuneo
  - SAPIENZA UNIVERSIT DI ROMA - POLO PONTINO - OSPEDALE S. MARIA GORETTI LATINA - UOC Ematologia, Latina
  - OSPEDALE VITO FAZZI LECCE - Hematologia, Lecce
  - OSPEDALE SAN RAFFAELE - Unità di Ricerca Clinica Linfomi Dipartimento di Onco-ematologia, Milan
  - AZIENDA OSPEDALIERO UNIVERITARIA DI MODENA - Ematologia, Modena
  - POLICLINICO SAN MATTEO - SC Ematologia, Pavia
  - OSPEDALE S. MARIA DELLE CROCI - Dipartimento di Oncologia ed Ematologia, Ravenna
  - AOU CITTA DELLA SALUTE E DELLA SCIENZA DI TORINO - Ematologia, Torino
  - OSPEDALE MAGGIORE ASUGI - UCO Ematologia, Trieste
- INSTITUTO PORTUGUES DE ONCOLOGIA DE LISBOA FRANCISCO GENTIL - Departamento Hematologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No